CLINICAL TRIAL: NCT04038190
Title: A Cluster-randomized Trial of a Behavioral Activation Intervention Administered in a College Freshman Orientation Course
Brief Title: A Behavioral Activation Intervention Administered in a College Freshman Orientation Course
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Kansas (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00143954; 1R01AA027791-01 (NIH)
Record Dates: First submitted 2019-06-27; First posted 2019-07-30 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Alcohol; Use, Problem; Stress; Binge Eating; Depression
Keywords: behavioral activation; prevention; reinforcement; college students
MeSH Terms: conditions — Alcoholism; Bulimia; Depression

STUDY DESIGN:
Intervention Model Description: The purpose of the study is to conduct a cluster randomized trial testing BA administered in a semester-long (16 week) freshman orientation course, compared to a standard orientation course in 540 freshmen spread over 36 course sections (18 sections each of the BA and standard orientation format). A 5-month post-treatment assessment will measure durability of effects. Mediation analyses will test mechanisms of action. A random sample of 20% of participants will complete a 17 month follow up to examine long term effects.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Activation Course (Experimental): Behavioral activation course condition administered in a college freshman orientation seminar
  Interventions: Behavioral: behavioral activation
- Standard Orientation Course (No Intervention): Standard freshman orientation seminar course condition

INTERVENTIONS:
Behavioral: behavioral activation — Behavioral activation (BA) is an intervention that indirectly addresses psychopathy by guiding individuals to identify goals in their lives, and encouraging individuals to engage in reinforcing activities that align with their goals (Lejuez et al, 2001). While initially used to treat depression, BA has been efficaciously applied to substance use because BA acts on the same reinforcement system common to many disorders (Daughters et al., 2018).
  Arms: Behavioral Activation Course

SUMMARY:
The transition from high school to college is a developmentally sensitive period that is high risk for escalations in alcohol use. Although risky drinking is a common problem among freshmen, engagement in treatment services is very low. The proposed study will test a behavioral activation intervention that addresses factors limiting participation in standard treatment services by targeting alcohol use indirectly, by directly addressing concerns most relevant to incoming college freshmen, and by integrating an intervention into the college curriculum.

DETAILED DESCRIPTION:
The transition from high school to college is a developmentally sensitive period that is high risk for escalations in alcohol use. Although risky drinking is a common problem among freshmen, engagement in treatment services is very low. Low rates of engagement with treatment resources may occur because interventions target drinking directly at a time when students may be uninterested in changing their drinking. Moreover, with a targeted focus on alcohol use, current interventions also do not address the concerns of incoming freshmen, such as stress and sleep. Approaches that address the problems students are most concerned about, that also indirectly reduce drinking, may be particularly effective.

Behavioral activation (BA) is an intervention that indirectly addresses psychopathy by guiding individuals to identify goals in their lives, and encouraging individuals to engage in reinforcing activities that align with their goals (Lejuez et al, 2001). While initially used to treat depression, BA has been efficaciously applied to substance use because BA acts on the same reinforcement process implicated in problem drinking. BA addresses drinking without specific reference to alcohol use by focusing on engagement in reinforcing activities that align with students' goals. A pilot study provided initial indication that a brief BA intervention administered in a semester-long freshman orientation course resulted in a significant decrease in drinking-related problems, compared to standard orientation (Reynolds et al. 2011). Notably, the approach never raised the issue of drinking unless raised by a student themselves.

The purpose of the study is to conduct a fully powered cluster randomized trial testing BA administered in a semester-long (16 week) freshman orientation course, compared to a standard orientation course in 540 freshmen spread over 36 course sections (18 sections each of the BA and standard orientation format). A 5-month post-treatment assessment will measure durability of effects. Mediation analyses will test mechanisms of action and moderation analyses will examine factors related to efficacy. A random sample of 20% of participants will complete a 17 month follow up, which will occur at the end of their sophomore year of college, to examine long term effects. With this proposed R01, the investigators will test a promising intervention with BA that addresses factors limiting participation in other programs by not targeting alcohol directly and by integrating an intervention into college curriculum, with the additional benefit of testing mediators to guide future work. This application represents a first step toward developing an intervention course that could be widely disseminated to address the persistent college drinking problem and its many consequences.

ELIGIBILITY:
Inclusion Criteria:

* College freshmen enrolled in UNIV 101 freshman seminar courses at the University of Kansas assigned to the study

Exclusion Criteria:

* None

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
alcohol consumption | baseline, 2 months, 4 months, and 8 months; 17 months for participants in Years 1-2
  Alcohol-Use Disorders Identification Test- Consumption Questions (AUDIT-C), which are the first three items of the AUDIT 10-item measure that asses frequency of drinking, typical quantity, and frequency of heavy drinking occasions (Saunders et al, 1993; Bush et al, 1998; DeMartini et al 2012). Responses are on a likert scale ranging from 0-4. The 3 items are summed for a total score with a possible range of 0-12, with higher scores indicating riskier drinking behavior.
high-intensity drinking (2+ times in excess of NIAAA low risk drinking guidelines for males and females) | baseline, 2 months, 4 months, and 8 months; 17 months for participants in Years 1-2
  The 30-day Time Line Follow Back-Computerized (TLFB-C) assessment will be used to measure alcohol consumption in the past 30 days (Sobell et al, 1996; Sobell & Sobell, 1992; Sobell & Sobell, 2008). The measure will be used to obtain the frequency at which individuals engaged in high-intensity drinking of 8+ drinks for males or 10+ drinks for females in one occasion.
alcohol-related problems | baseline, 2 months, 4 months, and 8 months; 17 months for participants in Years 1-2
  Alcohol-Use Disorders Identification Test- Problem Questions (AUDIT-P) are the last 7 items of the full AUDIT that assess increased salience of drinking, morning drinking, guilt after drinking, blackouts, alcohol-related injuries, and drinking that others are concerned about (Saunders et al, 1993; O'Hare & Sherrer, 2005). Responses are on a likert scale ranging from 0-4. The 7 items are summed for a total score with a possible range of 0-28, with higher scores indicating greater alcohol-related problems.
exceeding clinical cutoff of 8+ for hazardous/harmful drinking | baseline, 2 months, 4 months, and 8 months; 17 months for participants in Years 1-2
  The Alcohol-Use Disorders Identification Test (AUDIT) is designed to assess hazardous alcohol use and alcohol-related problems. The AUDIT has 10 items that assesses frequency of drinking, typical quantity, frequency of heavy drinking, impaired control over drinking, increased salience of drinking, morning drinking, guilt after drinking, blackouts, alcohol-related injuries, and others concerned about (Saunders et al, 1993). Responses are on a likert scale ranging from 0-4. The 10 items are summed for a total score with a possible range of 0-40, with higher scores indicating greater likelihood of hazardous drinking behavior.

SECONDARY OUTCOMES:
depression | baseline, 2 months, 4 months, and 8 months; 17 months for participants in Years 1-2
  Depression will be measured using the Depression Anxiety Stress Scale (DASS-21), a 21 item measure designed to assess depression, anxiety and stress (Lovibond & Lovibond, 1995). The measure provides scales for depression, anxiety, and stress and conceptualizes the difference between normal and clinical populations as a matter of degree. Thus, the DASS-21 is appropriate for use in a non-clinical, college sample. The depression scale assesses dysphoria, hopelessness, devaluation of life, self-deprecation, lack of interest / involvement, anhedonia and inertia with 7 items. Items are on a 4-point Likert scale ranging from 0-3 and can be summed for a scale score ranging from 0-21. Higher scores indicate more depression.
binge eating | baseline, 2 months, 4 months, and 8 months; 17 months for participants in Years 1-2
  Binge eating will be measured with the Eating Pathology Symptoms Inventory (EPSI; Forbush et al., 2013). The EPSI conceptualizes eating behavior on a dimensional scale and is appropriate for use in samples with and without eating disorders. The binge eating subscale will be used in the proposed study, which includes items on overeating and loss of control eating. The binge eating subscale has 8 items with Likert scale responses from 0=never to 4= very often. Items are summed for a scale score ranging from 0-32. Higher scores indicate more frequent experiences with binge eating behavior.
stress | baseline, 2 months, 4 months, and 8 months; 17 months for participants in Years 1-2
  Stress will be measured using the Depression Anxiety Stress Scale-21 (DASS-21), a 21 item measure designed to assess depression, anxiety and stress (Lovibond & Lovibond, 1995). The measure conceptualizes the difference between normal and clinical populations in stress as a matter of degree. Thus, the DASS-21 is appropriate for use in a non-clinical, college sample. b. The stress scale is sensitive to levels of chronic non-specific arousal. It assesses difficulty relaxing, nervous arousal, and being easily upset / agitated, irritable / over-reactive and impatient with 7 items. Items are on a 4-point Likert scale ranging from 0-3 and can be summed for a scale score ranging from 0-21. Higher scores indicate more stress.

OTHER OUTCOMES:
delay discounting | baseline, 2 months, 4 months, and 8 months; 17 months for participants in Years 1-2
  Delay Discounting will be measured using a titrating binary choice task, which uses hypothetical money rewards to assess the degree to which a reward is discounted due to delay. The magnitude of the delayed monetary amount will be $50 and $200 available after a specified delay (1 day, 1 wk, 1 month, 6 months, 1 yr, 5 yrs). Subjects will indicate if they prefer the immediate amount of money or the alternative with a mouse-click and the computerized algorithm will adjust the immediate reward over 6 trials to determine an indifference point for each amount/delay pairing. Indifference points will be used to calculate a delay-discount rate. Higher delay discount rates indicate strong discounting and a preference for immediate rewards.
reinforcement from alcohol-related and alcohol-free activities | baseline, 2 months, 4 months, and 8 months; 17 months for participants in Years 1-2
  The Adolescent Reinforcement Survey Schedule - Alcohol Use Version assesses the frequency of past-month engagement in and enjoyment derived from 45 activities (Hallgren et al, 2016). Each question is posed twice - once to assess the frequency and enjoyment of the activity while using alcohol and the once to assess the frequency and enjoyment of the activity while not using alcohol. Items range from 0-4. Frequency and enjoyment items are summed to form respective scores. From these scales, two subscales are created for alcohol-related reinforcement and alcohol-free reinforcement, calculated as the cross product between frequency and enjoyment items for alcohol-related and alcohol-free questions. The two subscales are used to calculate the outcome, the total reinforcement ratio (TRR) between alcohol-related and alcohol-free reinforcement. The ratio has values between 0 and 1, with higher values indicating more relative enjoyment of activities when using alcohol.
coping-motivated drinking | baseline, 2 months, 4 months, and 8 months; 17 months for participants in Years 1-2
  The Drinking Motives Questionnaire-Revised (DMQ-R) designed to measure the relative frequency of drinking for four distinct reason motives: enhancement, social, conformity, and coping (Cooper, 1994; Cox & Klinger, 1988). The measure produces four scales that correspond with the four motives. The present study will use the coping motives scale, which contains 5 items. Items are assessed on a Likert scale ranging from 1-5 and are summed for form a scale score, which higher scores indicating greater frequency in coping-motivated drinking.
grade point average (GPA) | baseline, 2 months, 4 months, and 8 months; 17 months for participants in Years 1-2
  Academic performance will be measured using participate grade point average (GPA).
alcohol violations on campus | baseline, 2 months, 4 months, and 8 months; 17 months for participants in Years 1-2
  Participants alcohol violations at the University of Kansas will be documented at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Tera L Fazzino, PhD, Principal Investigator — University of Kansas
Locations (1):
- University of Kansas, Lawrence, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fazzino TL, Kunkel A, Bellitti J, Romine RS, Yi R, McDaniel C, Lejuez CW. Engagement with Activity Monitoring During a Behavioral Activation Intervention: A Randomized Test of Monitoring Format and Qualitative Evaluation of Participant Experiences. Behav Change. 2023 Jun;40(2):103-116. doi: 10.1017/bec.2022.7. Epub 2022 Jun 16. PMID 37583941
- [Result] Fazzino TL, Lejuez CW, Yi R. A behavioral activation intervention administered in a 16-week freshman orientation course: Study protocol. Contemp Clin Trials. 2020 Mar;90:105950. doi: 10.1016/j.cct.2020.105950. Epub 2020 Jan 23. PMID 31982647
- [Result] Jun D, Fazzino TL. Associations between Alcohol-Free Sources of Reinforcement and the Frequency of Alcohol and Cannabis Co-Use among College Freshmen. Int J Environ Res Public Health. 2023 Feb 7;20(4):2884. doi: 10.3390/ijerph20042884. PMID 36833579